CLINICAL TRIAL: NCT06157268
Title: Trial Readiness and Trial Fitness for Congenital Myopathies: a 2-year Prospective Natural History Study Including a Cross-sectional Study on Muscle Fatigability
Brief Title: The Natural History and Muscle Fatigability of Patients With Congenital Myopathies.
Acronym: READYCOM
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: NL83069.000.23; W.OR22-10 (Other Grant/Funding Number: Prinses Beatrix Spierfonds)
Record Dates: First submitted 2023-11-09; First posted 2023-12-05 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Central Core Disease; Multi-Minicore Disease; Nemaline Myopathy; Centronuclear Myopathy
Keywords: Natural history study; Outcome measures; Congenital myopathy; Muscle disease
MeSH Terms: conditions — Myopathy, Central Core; Minicore Myopathy with External Ophthalmoplegia; Myopathies, Nemaline; Myopathies, Structural, Congenital; Myotonia Congenita; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Core myopathies: Patients with a genetically confirmed core myopathy
  Interventions: Other: Natural history and non therapeutical therapy
- Nemaline myopathy: Patients with a genetically confirmed nemaline myopathy
  Interventions: Other: Natural history and non therapeutical therapy
- Centronuclear myopathy: Patients with a genetically confirmed centronuclear myopathy
  Interventions: Other: Natural history and non therapeutical therapy

INTERVENTIONS:
Other: Natural history and non therapeutical therapy — This study concerns a natural history study part and a muscle fatigability part.
  For the natural history study no interventions will be used. For the muscle fatigability part non therapeutical therapies will be used. This includes endurance tests, isokinetic dynamometry and repetitive nerve stimulation.

SUMMARY:
Core myopathies (CCD/MmD), nemaline myopathies (NEM) and centronuclear myopathies (CNM) are three types of rare congenital myopathies. Not much is known about the natural history and no curative treatment is available for these groups. Also patients report fatigability as one of their symptoms. The goal of this observational study is to study the natural history during 24 months to achieve trial readiness and to study the muscle fatigability in CCD/MmD, NEM and CNM.

DETAILED DESCRIPTION:
Rationale: Patients with CCD/MmD, NEM and CNM report symptoms of weakness in the arms and legs. Other symptoms include weakness of the respiratory, facial and swallowing muscles. No treatments are available for congenital myopathies (CM) to slow down or cure the disease. A few type I-II trials have taken place and more are expected. Therefore it is important to reach trial readiness. To create trial readiness, there is a need for natural history study to create a detailed report of the disease course and a selection of the most sensitive clinical and functional outcome measures and biomarkers. Besides muscle weakness, several patients report muscle fatigability. This has not been investigated systematically in CM. The lack of evidence calls for a cross-sectional study assessing muscle fatigability and neuromuscular transmission in CM.

Objectives: i) To assess the natural disease course of CCD/MmD, NEM and CNM during 24 months. ii) To select relevant and sensitive clinical and functional outcome measures and biomarkers. iii) To assess the severity of muscle fatigability in CCD/MmD, NEM and CNM.

Study design: Patients with a genetically confirmed CCD/MmD, NEM or CNM will be able to participate in this study. The study consist of 2 parts. Part 1: a prospective cohort study with 5 visits every 6 months, for a total of 2 years. 45 patients will be included for this part. Part 2: an observational study with 2 visits. For this part 75 patients will be included. There will be an overlap in patients for the two parts. So a total of approximately 100 patients will be included. A large set of tests will be performed to assess the full capabilities of the patient, e.g. muscle strength/endurance, muscle imaging (MRI/ultrasound), activities, walking ability, quality of life, muscle fatigability and the feeling of fatigue.

ELIGIBILITY:
Inclusion Criteria for the natural history:

* 2 years or older
* Willing and able to complete the measurement protocol
* Willing and able to travel to Nijmegen and Utrecht
* Dutch-speaking
* Genetically-confirmed congenital myopathy (CCD/MmD, NEM, and CNM)

Inclusion Criteria for the fatigability study:

* 8-60 years old
* Willing and able to complete the measurement protocol
* Willing and able to travel to Nijmegen and Utrecht
* Dutch-speaking
* Genetically-confirmed congenital myopathy (CCD/MmD, NEM, and CNM)
* Willing to stop taking pyridostigmine and/or salbutamol 24 hours before the visit.

Exclusion Criteria for both parts:

Other neuromuscular, psychiatric or neurological disorders.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 45 patients will be included in the natural history study and 75 patients in the fatigability study, with some patients in both studies. The participants will be equally divided over three groups (CCD/MmD, NEM, CNM). Patients will be identified through patient databases of the Radboudumc and UMC Utrecht and patient groups. If more than 15/25 patients per group are willing to participate, we will select patients based on age and severity to have a good representation of the entire/complete disease spectrum.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change of Motor Function Measure (MFM) | Change from baseline at 6, 12, 18 and 24 months
  Global motor functioning. The main outcome is the change in MFM score over a period of 2 years. The scores of the patients will also be compared to reference values.
Endurance shuttle test - fatigability part | At assessment 1 or 2 of the fatigability part of the study. Which day is dependent on the preference of the patient and planning possibilities.
  Patients walk/move blocks/move pegs at a personalised set speed. The main outcome is if the patient drops out due to the speed being too low. If the patient drops out the time until dropout is noted.

SECONDARY OUTCOMES:
Change of 6-minute walk test (6MWT) (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  How far the patient can walk in 6 minutes. The first and last minute will be compared to each other.
Accelerometry - change of extent and intensity of physical activity in daily life (all ages) | Change from baseline at 6, 12, 18 and 24 months
  Physical activity in daily life will be assessed by wearing an wrist worn accelerometer (GENEActiv original devices) for 7 days.
Change of bone density (DEXA scan) (6 years and older) | Change from baseline at 24 months
  The bone density of the spine and hip will be measured by a DEXA scan.
Change of graded and timed rise from floor (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  The time it takes to rise from the floor
Handheld dynamometry (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Maximal voluntary isometric contraction will be measured by handheld dynamometry (m. biceps brachii, m. quadriceps, grip strength, all bilaterally)
Creatine Kinase | At baseline
  Blood level of Creatine Kinase
Vitamin D3 | At baseline
  Blood level of Vitamin D3
Calcium | At baseline
  Blood level of calcium
Liver function panel | At baseline
  Blood level of bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, gamma-glutamyltransferase GGT, albumin, bile acids and full blood count.
Manual muscle testing (MMT) (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Muscle power of individual muscle groups can be assessed by muscle power measurements and graded in correspondence with the Medical Research Council (MRC) scale.
Change in muscle fattening by quantitative lower extremity muscle MRI (10 years and older) | Change from baseline at 24 months
  A lower extremity muscle MRI will be performed in participants who are able to lie supine and still for 20 minutes and who are not dependent on respiratory equipment. Muscle fattening will be assessed by Regions of Interest (ROIs) (quantitative) and modified Mercuri score (semi-quantitative).
Change of muscle atrophy by quantitative lower extremity muscle MRI (10 years and older) | Change from baseline at 24 months
  A lower extremity muscle MRI will be performed in participants who are able to lie supine and still for 20 minutes and who are not dependent on respiratory equipment. Atrophy will be assessed by muscle volume score (semi-quantitative).
Change in muscle atrophy (cm) assessed by muscle ultrasound (all ages) | Change from baseline at 24 months
  Muscle atrophy of the leg, arm, back, abdominal muscles and diaphragm will be assessed by muscle ultrasound.
Change in muscle fattening (echo-intensity) assessed by muscle ultrasound (all ages) | Change from baseline at 24 months
  Muscle fattening of the leg, arm, back, abdominal muscles and diaphragm will be assessed by muscle ultrasound.
Range of motion (all ages) | Change from baseline at 6, 12, 18 and 24 months
  The range of motion of the elbows, fingers, knees and ankles is noted bilaterally by goniometry.
Pulmonary function - change of forced vital capacity (percentage predicted) (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Obtained with handheld spirometry in sit and supine.
Pulmonary function - change of forced expiratory volume in the first second (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Obtained with handheld spirometry in sit and supine.
Pulmonary function - change of maximal expiratory pressure (cmH2O) (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Obtained with handheld device.
Pulmonary function - change of maximal inspiratory pressure (cmH2O) (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Obtained with handheld device.
Pulmonary function - change of sniff nasal inspiratory pressure (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Obtained with handheld device.
Vignos and Brooke scale (all ages) | Change from baseline at 6, 12, 18 and 24 months
  The Brooke (score 1-6) and Vignos (score 1-10) scales provide ordinal data to assess the upper and lower extremity functions. A lower score indicates more functionality.
Isokinetic dynamometry (quadriceps and hamstrings or biceps and triceps) (8-60 years old) - fatigability part | At assessment 1 or 2 of the fatigability part of the study. Which day is dependent on the preference of the patient and planning possibilities.
  Peak torque, time to peak torque, change in torque from first third to last third, acceleration time and deceleration time for 3, 5 and 30 repetitions at a set speed. For the 30 repetitions how many repetitions until failure is also noted.
Change in surface electromyography (EMG) amplitude and median frequency during isokinetic dynamometry with surface EMG (quadriceps and hamstrings or biceps and triceps) (8-60 years old) - fatigability part | At assessment 1 or 2 of the fatigability part of the study. Which day is dependent on the preference of the patient and planning possibilities.
  On the quadriceps/hamstrings or biceps/triceps surface EMG amplitude and median frequency will be measured.
Repetitive nerve stimulation (RNS) (8-60 years old) - fatigability part | At assessment 1 or 2 of the fatigability part of the study. Which day is dependent on the preference of the patient and planning possibilities.
  We will stimulate the n. ulnaris, n. accesorius and n. facialis at 3 Hz to measure the m abductor digiti minimi, m. trapezius and m nasalis. The decrement/increment will be determined by the compound muscle action potential amplitude and area.
  The RNS will be performed before and after 60 seconds of voluntary contraction.
Checklist individual strength (CIS) questionnaire fatigue subscale (18 years and older) | Change from baseline at 6, 12, 18 and 24 months
  The CIS is a questionnaire rating four subscales: subjective tiredness, concentration, motivation and physical activity. It consists of 20 items on a 7-point scale. We will use the Fatigue subscale. A CIS fatigue scale ≥ 35 points to severe fatigue.
Fatigue severity scale questionnaire (12 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Nine-questions scale about the impact of fatigue on the patient's life. Each item is scored on a 7 point scale. A higher score indicates greater fatigue/greater impact of fatigue on daily life.
PedsQL multidimensional fatigue scale (MFS) (2-17 years old) | Change from baseline at 6, 12, 18 and 24 months
  The PedsQL MFS assesses subjective fatigue in three domains with 6 items each, namely General Fatigue Scale, Sleep/Rest Fatigue Scale, and Cognitive Fatigue Scale. Each item is scored on a three point scale ranging from not at all to a lot for children aged 5-7 and a five point scale from never to almost always for the others. Higher scores indicates less symptoms.
PROMIS Fatigue Short Form questionnaire (all ages) | Change from baseline at 6, 12, 18 and 24 months
  Consists of 8 items representing the most informative items from the PROMIS item bank. The PROMIS Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. For patients younger than 18 a parent proxy is also available. The items are scored form 1-5 with a higher score indicating more fatigue.
McGill pain questionnaire (MPQ) (12 years and older) | Change from baseline at 6, 12, 18 and 24 months
  The MPQ consists of 4 components: a pain word list to state the type and intensity of the pain, questions about the effect on daily life, a visual-analogue scale for pain intensity and questions about the location and course of the pain.
Wong-Baker Faces Pain Scale (2-11 years old) | Change from baseline at 6, 12, 18 and 24 months
  The Wong-Baker Faces Pain Scale was originally created for children to help them communicate about their pain. It has six types of faces ranging from no hurt (0) tot hurts worst (10).
PedsQL generic quality of life (2-17 years old) | Change from baseline at 6, 12, 18 and 24 months
  The PedsQL generic quality of life questionnaire consists of 8 items on physical functioning, 5 items on emotional functioning, 5 items on social functioning, and 5 items on school functioning. Each item is scored on a 0-4 scale. The items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate a better outcome.
Short Form 36 (SF36) quality of life scale (18 years and older) | Change from baseline at 6, 12, 18 and 24 months
  The adult Quality of Life is measured by the SF36/RAND36 questionnaire. The SF36/RAND36 addresses eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. It has a total of 36 items.
Activlim questionnaire (7-17 years old) | Change from baseline at 6, 12, 18 and 24 months
  ACTIVLIM assesses the ability to perform 22 activities of daily life on a 3-point scale from impossible to easy. The questionnaires will be answered by the parents of the patient.
Impact on participation and autonomy (18 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Questionnaire about participation and autonomy in daily life with 41 questions on a ordinal 3- or 5-point likert scale. Higher scores indicate more obstacles in participation and autonomy.
Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P) (18 years and older) | Change from baseline at 6, 12, 18 and 24 months
  USER-P Restrictions scale is a patients-reported outcome measures with 32 questions focusing on daily activities including school and work. Each item is scored on a 4-, 5-, and 6-point Likert scale. A higher score indicates more participation.
Borg rating scale of perceived exertion (5 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Borg Rating Scale of Perceived Exertion is a way of measuring physical activity intensity level. Perceived exertion is based on the physical sensations a person experiences during physical activity. It is scored 6-20 with a higher score indicating a greater perceived exertion.
  Participants will be asked to score the intensity level at the beginning and at the end of the 6MWT.
Hospital anxiety and depression scale (18 years and older) | Change from baseline at 6, 12, 18 and 24 months
  Questionnaire about the main complaints of anxiety and depression with 7 items each on a 4-point Likert scale. A higher score indicates more complaints.
PedsQL neuromuscular module (NMM) (2-17 years old) | Change from baseline at 6, 12, 18 and 24 months
  The PedsQL NMM questionnaire consists of 25 questions in three domains: Neuromuscular disease, communication and family resources. Each item is scored on a 0-4 scale. The items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate a better outcome.
Resilience evaluation scale (18 years and older) | Change from baseline at 6, 12, 18 and 24 months
  9-Item questionnaire on psychological resilience with each item being scored from 0-4, higher scores indicating greater resilience.
Effects of pyridostigmine and/or salbutamol (8-60 years old) - fatigability part | At baseline of the fatigability part of the study
  We will ask patients if they use pyridostigmine and/or salbutamol. If they use it we will ask how often, what the effects are and how long those effects last.

CONTACTS AND LOCATIONS:
Overall Officials: Nicol Voermans, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
Research data is open access shared upon publication, provided that this complies with privacy regulations. The Donders Repository is the default repository for sharing the investigators' data.